CLINICAL TRIAL: NCT02886897
Title: A Phase II Study of Combinations of Dendritic Cells and Cytokine-induced Killer Cell （D-CIK) Immunotherapy And Anti-Programmed Death-1 In Refractory Solid Tumors
Brief Title: A Study of Combinations of D-CIK Immunotherapy And Anti-PD-1 In Refractory Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jianchuan Xia, Director of Biotherapy;Principal Investigator;Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2016-036-01
Record Dates: First submitted 2016-08-14; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Hepatocellular Carcinoma; Renal Cell Carcinoma; Bladder Cancer; Colorectal Cancer; Non-small-cell Lung Cancer; Breast Cancer
Keywords: Refractory solid tumors; Dendritic and Cytokine-induced killer cell; Anti-PD-1 antibody; Combination immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- D-CIK and anti-PD-1 Immunotherapy (Experimental): D-CIK was incubated with anti-PD-1 antibody before infused back into participants
  Interventions: Biological: D-CIK and anti-PD-1 antibody

INTERVENTIONS:
Biological: D-CIK and anti-PD-1 antibody — Autologous dendritic and cytokine-induced killer cells (D-CIK)(1.0-1.5*10^10 cells)were incubated with anti-PD-1 antibody and infused into participants.

SUMMARY:
Background: Combinations of dendritic and cytokine-induced killer cell (D-CIK) based adoptive immunotherapy and anti-PD-1 antibody may enhance the immune response and stop cancer cells from growing.

Objective: Phase II clinical trial to investigate the safety, clinical activity and toxicity of combinations of D-CIK and anti-PD-1 antibody in patients with treatment-refractory solid tumors.

Methodology: Phase II clinical trial in patients with advanced metastatic hepatocellular carcinoma, renal cell carcinoma,bladder cancer,colorectal cancer,non-small-cell lung cancer,breast cancer and other solid cancers. The D-CIK was isolated from peripheral blood of participants,then activated,expanded and incubated with anti-PD-1 antibody before infusion. The enough number (1.0-1.5 *10^10 cells) of D-CIK were infused back into participants.

DETAILED DESCRIPTION:
Heparinized peripheral blood was obtained from participants over a 2-week period. PBMCs were separated by Ficoll-Hypaque gradient centrifugation, suspended in X-VIVO 15 serum-free medium, and culture with 1000 U/ml rhIFN-γfor the first 24 h, followed by stimulation with 100 ng/ml OKT3 , 1000 U/ml rhIL-2 and 100 U/ml IL-1α to activate the CIK.Dendritic cells were incubated with CIK. Fresh medium containing 1000 U/ml rhIL-2 was added every 2 days and the cell density was maintained at 2×10^6 cells/mL.D-CIK were harvested, washed, and resuspended after culture for 14 days. Before cell transfer,D-CIK were incubated with anti-PD-1 antibody,and a fraction of the D-CIK were collected to assess their number, phenotype, and viability of cells, and to test for possible contamination by bacteria, fungi, or endotoxins. Then, autologous D-CIK (1.0-1.5*10^10 cells) were transferred to patients via intravenous infusion. Generally, participants received at least 4 cycles of treatment at 2-week intervals or received doses until disease progression occurred. If the participants were disease-stable, additional cycles of maintenance treatment were eligible.

Participants will be evaluated for the safety, clinical activity and toxicity. The primary end point was the objective response for each participant at the time of D-CIK and anti-PD-1 infusion as assessed by RECIST. Peripheral blood of patients were also assessed for related cytokine using ELISPOT assays. Additional,the investigators will evaluate tumor markers in participants with clinical response/non-response by immunohistochemical staining of tumor sections from previous diagnostic or therapeutic biopsy samples to determine the predictive biomarker that may be used in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Participantswith treatment-refractory advanced hepatocellular carcinoma, renal cell carcinoma,bladder cancer,colorectal cancer,non-small-cell lung cancer,breast cancer and other solid cancers.
* Age 18 to 75 years.
* Willing to sign a durable power of attorney.
* Able to understand and sign the Informed Consent Document.
* Life expectancy of greater than three months.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the preparative regimen.
* Adequate organ function.
* Serology:

  * Seronegative for HIV antibody.
  * Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
* Hematology:

  * WBC (> 3000/mm(3)).
  * Platelet count greater than 100,000/mm(3).
  * Hemoglobin greater than 8.0 g/dl.
* Chemistry:

  * Serum ALT/AST less or equal to 2.5 times the upper limit of normal.
  * Serum creatinine less than or equal to 1.6 mg/dl.
  * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.

Exclusion Criteria:

* Previous treatment with anti-CTLA-4 and anti-PD-1/PD-L1.
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* History of autoimmune disease
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Concurrent antineoplastic therapies and systemic steroid therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival(PFS) | 12 Months
  PFS is defined as the time from the combined therapy until objective tumor progression or death.

SECONDARY OUTCOMES:
Overall survival (OS) | 12 Months
  OS is defined as the time from the combined therapy until death from any cause
Laboratory findings | 6 Months
  The number and secreted cytokines of CD3+ (or CD8+ or CD4+ or CD56+) T cells
Objective response rate | 12 Months
  The total number of Complete remission and Partial remission (According to the response criteria in solid tumor(RECIST))
Severity of adverse events | 12 Months
  According to National Cancer Institute Common Terminology Criteria for Adverse Events（NCI-CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Xin Zeng, Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University, Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Taube JM, Anders RA, Young GD, Xu H, Sharma R, McMiller TL, Chen S, Klein AP, Pardoll DM, Topalian SL, Chen L. Colocalization of inflammatory response with B7-h1 expression in human melanocytic lesions supports an adaptive resistance mechanism of immune escape. Sci Transl Med. 2012 Mar 28;4(127):127ra37. doi: 10.1126/scitranslmed.3003689. PMID 22461641
- [Result] Lee JH, Lee JH, Lim YS, Yeon JE, Song TJ, Yu SJ, Gwak GY, Kim KM, Kim YJ, Lee JW, Yoon JH. Adjuvant immunotherapy with autologous cytokine-induced killer cells for hepatocellular carcinoma. Gastroenterology. 2015 Jun;148(7):1383-91.e6. doi: 10.1053/j.gastro.2015.02.055. Epub 2015 Mar 4. PMID 25747273
- [Result] Mahoney KM, Rennert PD, Freeman GJ. Combination cancer immunotherapy and new immunomodulatory targets. Nat Rev Drug Discov. 2015 Aug;14(8):561-84. doi: 10.1038/nrd4591. PMID 26228759
- [Result] Pan K, Guan XX, Li YQ, Zhao JJ, Li JJ, Qiu HJ, Weng DS, Wang QJ, Liu Q, Huang LX, He J, Chen SP, Ke ML, Zeng YX, Xia JC. Clinical activity of adjuvant cytokine-induced killer cell immunotherapy in patients with post-mastectomy triple-negative breast cancer. Clin Cancer Res. 2014 Jun 1;20(11):3003-11. doi: 10.1158/1078-0432.CCR-14-0082. Epub 2014 Mar 25. PMID 24668644
- [Result] Dai C, Lin F, Geng R, Ge X, Tang W, Chang J, Wu Z, Liu X, Lin Y, Zhang Z, Li J. Implication of combined PD-L1/PD-1 blockade with cytokine-induced killer cells as a synergistic immunotherapy for gastrointestinal cancer. Oncotarget. 2016 Mar 1;7(9):10332-44. doi: 10.18632/oncotarget.7243. PMID 26871284